CLINICAL TRIAL: NCT00730847
Title: A Post-marketing Surveillance (PMS) Study to Monitor the Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) Vaccine (Cervarix) in 3,000 Healthy Female Filipino Subjects When Administered According to the Prescribing Information From the Age of 10 Years Onwards.
Brief Title: A Study to Assess the Safety and Reactogenicity of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV) Vaccine (Cervarix) in Healthy Female Filipino Subjects Vaccinated According to the Prescribing Information From the Age of 10 Years Onwards.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: GSK received exemption from PDFDA on conduct of this post-marketing surveillance (PMS) study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 108160; 2017-000458-20 (EudraCT Number)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Human Papillomavirus Infection Leading to Cervical Cancer
Keywords: Cervarix; Filipinos; Safety and reactogenicity; Human papillomavirus
MeSH Terms: interventions — human papillomavirus vaccine, L1 type 16, 18

ARMS (1):
- Cervarix Group (Experimental): Healthy female subjects who received three doses of the Cervarix vaccine, administered intramuscularly in the deltoid region according to a 0, 1 and 6-month schedule.
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Cervarix — Three doses of Cervarix administered intramuscularly in the deltoid region, according to a 0, 1, 6-month vaccination schedule.
  Other Names: HPV-16/18 VLP/AS04 vaccine

SUMMARY:
The purpose of this study was to assess the safety and reactogenicity of GSK Biologicals' Cervarix vaccine in healthy female Filipino subjects from the age of 10 years onwards, as per the Bureau of Food and Drugs Directive of Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their LAR's can and will comply with the requirements of the protocol should be enrolled in the study.
* A female 10 years of age and above at the time of the first vaccination.
* Written informed consent obtained from the subject. For subjects below the legal age of consent, written informed consent must be obtained from the parent or legal guardian (legally acceptable representative -LAR) of the subject and informed assent must be obtained from the subject.
* Free of obvious health problems as established by medical history and history-directed physical examination before entering into the study.
* Subjects of childbearing potential must not be pregnant.
* Subjects must be of non-childbearing potential, or if the subject is of childbearing potential, she must be abstinent (and if so, this must be documented in the source documents at each vaccination visit) or must be using adequate contraception for 30 days prior to vaccination and continue for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or non-investigational product (pharmaceutical product or device).
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive prevention during the study period and up to two months after the last vaccine dose.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccine.
* Hypersensitivity to latex (found in syringe-tip cap and plunger).
* Known acute or chronic, clinically significant neurologic, haematological, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* Cancer or autoimmune disease under treatment.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study.
* Acute disease at the time of enrolment.

Min Age: 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2008-09-17 (Actual); Primary Completion 2012-01-16 (Actual); Study Completion 2012-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Philippines (2):
  - GSK Investigational Site, Ermita, Manila
  - GSK Investigational Site, Makati City

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=107921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Since this was a post-marketing study (PMS), subjects may have received one or two doses of Cervarix outside of the PMS.
Pre-assignment Details: Out of 743 subjects enrolled in the study, only 596 subjects received study vaccination.
  The whole set of data was not cleaned for this study. Analysis was performed on subjects with cleaned data and on subjects with missing data or unresolved data queries, or both. The overall group includes both cleaned and not cleaned data.
Groups:
- Cervarix Group: Healthy female subjects who received three doses of Cervarix vaccine administered intramuscularly in the deltoid region according to a 0, 1 and 6-month schedule.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 596
Completed | 465
Not Completed | 131
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 67
Not completed — Unknown completion status | 21
Not completed — Other | 24

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 596
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.8 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 596
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  South Asian | 594
  Chinese | 1
  Not specified | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity grade. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness and swelling above 50 millimeters (mm).
Time Frame: During the 7-day follow-up period (Days 0-6) after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and had the symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 578
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 576
  Any Pain, Dose 1 | 402
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 576
  Grade 3 Pain, Dose 1 | 25
  Any Redness, Dose 1: number analyzed (Participants) | 576
  Any Redness, Dose 1 | 116
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 576
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 576
  Any Swelling, Dose 1 | 76
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 576
  Grade 3 Swelling, Dose 1 | 3
  Any Pain, Dose 2: number analyzed (Participants) | 531
  Any Pain, Dose 2 | 309
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 531
  Grade 3 Pain, Dose 2 | 16
  Any Redness, Dose 2: number analyzed (Participants) | 531
  Any Redness, Dose 2 | 106
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 531
  Grade 3 Redness, Dose 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 531
  Any Swelling, Dose 2 | 60
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 531
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 482
  Any Pain, Dose 3 | 211
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 482
  Grade 3 Pain, Dose 3 | 7
  Any Redness, Dose 3: number analyzed (Participants) | 482
  Any Redness, Dose 3 | 69
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 482
  Grade 3 Redness, Dose 3 | 2
  Any Swelling, Dose 3: number analyzed (Participants) | 482
  Any Swelling, Dose 3 | 47
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 482
  Grade 3 Swelling, Dose 3 | 1
  Any Pain, Across doses | 430
  Grade 3 Pain, Across doses | 38
  Any Redness, Across doses | 168
  Grade 3 Redness, Across doses | 2
  Any Swelling, Across doses | 119
  Grade 3 Swelling, Across doses | 4

2. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, fever, gastrointestinal, headache, myalgia, rash and urticaria. Any fever = axillary temperature ≥ 37.5 degrees Celsius (°C). For other symptoms: Any = any solicited general symptom reported irrespective of intensity and relationship to study vaccination. Related = symptoms considered by the investigator as causally related to study vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 urticaria = urticaria distributed on at least 4 body areas. Grade 3 fever = axillary temperature > 39.0°C.
Time Frame: During the 7-day follow-up period (Days 0-6) after each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 576
Participants
  Any Arthralgia, Dose 1: number analyzed (Participants) | 575
  Any Arthralgia, Dose 1 | 76
  Grade 3 Arthralgia, Dose 1: number analyzed (Participants) | 575
  Grade 3 Arthralgia, Dose 1 | 2
  Related Arthralgia, Dose 1: number analyzed (Participants) | 575
  Related Arthralgia, Dose 1 | 35
  Any Fatigue, Dose 1: number analyzed (Participants) | 575
  Any Fatigue, Dose 1 | 120
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 575
  Grade 3 Fatigue, Dose 1 | 4
  Related Fatigue, Dose 1: number analyzed (Participants) | 575
  Related Fatigue, Dose 1 | 53
  Any Fever, Dose 1: number analyzed (Participants) | 575
  Any Fever, Dose 1 | 17
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 575
  Grade 3 Fever, Dose 1 | 1
  Related Fever, Dose 1: number analyzed (Participants) | 575
  Related Fever, Dose 1 | 7
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 575
  Any Gastrointestinal, Dose 1 | 46
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 575
  Grade 3 Gastrointestinal, Dose 1 | 3
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 575
  Related Gastrointestinal, Dose 1 | 10
  Any Headache, Dose 1: number analyzed (Participants) | 575
  Any Headache, Dose 1 | 90
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 575
  Grade 3 Headache, Dose 1 | 3
  Related Headache, Dose 1: number analyzed (Participants) | 575
  Related Headache, Dose 1 | 29
  Any Myalgia, Dose 1: number analyzed (Participants) | 575
  Any Myalgia, Dose 1 | 91
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 575
  Grade 3 Myalgia, Dose 1 | 4
  Related Myalgia, Dose 1: number analyzed (Participants) | 575
  Related Myalgia, Dose 1 | 39
  Any Rash, Dose 1: number analyzed (Participants) | 575
  Any Rash, Dose 1 | 9
  Grade 3 Rash, Dose 1: number analyzed (Participants) | 575
  Grade 3 Rash, Dose 1 | 0
  Related Rash, Dose 1: number analyzed (Participants) | 575
  Related Rash, Dose 1 | 4
  Any Urticaria, Dose 1: number analyzed (Participants) | 575
  Any Urticaria, Dose 1 | 8
  Grade 3 Urticaria, Dose 1: number analyzed (Participants) | 575
  Grade 3 Urticaria, Dose 1 | 0
  Related Urticaria, Dose 1: number analyzed (Participants) | 575
  Related Urticaria, Dose 1 | 3
  Any Arthralgia, Dose 2: number analyzed (Participants) | 529
  Any Arthralgia, Dose 2 | 43
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 529
  Grade 3 Arthralgia, Dose 2 | 1
  Related Arthralgia, Dose 2: number analyzed (Participants) | 529
  Related Arthralgia, Dose 2 | 15
  Any Fatigue, Dose 2: number analyzed (Participants) | 529
  Any Fatigue, Dose 2 | 81
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 529
  Grade 3 Fatigue, Dose 2 | 6
  Related Fatigue, Dose 2: number analyzed (Participants) | 529
  Related Fatigue, Dose 2 | 35
  Any Fever, Dose 2: number analyzed (Participants) | 529
  Any Fever, Dose 2 | 11
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 529
  Grade 3 Fever, Dose 2 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 529
  Related Fever, Dose 2 | 9
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 529
  Any Gastrointestinal, Dose 2 | 32
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 529
  Grade 3 Gastrointestinal, Dose 2 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 529
  Related Gastrointestinal, Dose 2 | 9
  Any Headache, Dose 2: number analyzed (Participants) | 529
  Any Headache, Dose 2 | 55
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 529
  Grade 3 Headache, Dose 2 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 529
  Related Headache, Dose 2 | 20
  Any Myalgia, Dose 2: number analyzed (Participants) | 529
  Any Myalgia, Dose 2 | 52
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 529
  Grade 3 Myalgia, Dose 2 | 2
  Related Myalgia, Dose 2: number analyzed (Participants) | 529
  Related Myalgia, Dose 2 | 20
  Any Rash, Dose 2: number analyzed (Participants) | 529
  Any Rash, Dose 2 | 7
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 529
  Grade 3 Rash, Dose 2 | 1
  Related Rash, Dose 2: number analyzed (Participants) | 529
  Related Rash, Dose 2 | 3
  Any Urticaria, Dose 2: number analyzed (Participants) | 529
  Any Urticaria, Dose 2 | 6
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 529
  Grade 3 Urticaria, Dose 2 | 1
  Related Urticaria, Dose 2: number analyzed (Participants) | 529
  Related Urticaria, Dose 2 | 1
  Any Arthralgia, Dose 3: number analyzed (Participants) | 481
  Any Arthralgia, Dose 3 | 30
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 481
  Grade 3 Arthralgia, Dose 3 | 3
  Related Arthralgia, Dose 3: number analyzed (Participants) | 481
  Related Arthralgia, Dose 3 | 13
  Any Fatigue, Dose 3: number analyzed (Participants) | 481
  Any Fatigue, Dose 3 | 57
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 481
  Grade 3 Fatigue, Dose 3 | 3
  Related Fatigue, Dose 3: number analyzed (Participants) | 481
  Related Fatigue, Dose 3 | 28
  Any Fever, Dose 3: number analyzed (Participants) | 481
  Any Fever, Dose 3 | 12
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 481
  Grade 3 Fever, Dose 3 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 481
  Related Fever, Dose 3 | 8
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 481
  Any Gastrointestinal, Dose 3 | 15
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 481
  Grade 3 Gastrointestinal, Dose 3 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 481
  Related Gastrointestinal, Dose 3 | 6
  Any Headache, Dose 3: number analyzed (Participants) | 481
  Any Headache, Dose 3 | 39
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 481
  Grade 3 Headache, Dose 3 | 2
  Related Headache, Dose 3: number analyzed (Participants) | 481
  Related Headache, Dose 3 | 13
  Any Myalgia, Dose 3: number analyzed (Participants) | 481
  Any Myalgia, Dose 3 | 30
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 481
  Grade 3 Myalgia, Dose 3 | 1
  Related Myalgia, Dose 3: number analyzed (Participants) | 481
  Related Myalgia, Dose 3 | 13
  Any Rash, Dose 3: number analyzed (Participants) | 481
  Any Rash, Dose 3 | 4
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 481
  Grade 3 Rash, Dose 3 | 1
  Related Rash, Dose 3: number analyzed (Participants) | 481
  Related Rash, Dose 3 | 2
  Any Urticaria, Dose 3: number analyzed (Participants) | 481
  Any Urticaria, Dose 3 | 2
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 481
  Grade 3 Urticaria, Dose 3 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 481
  Related Urticaria, Dose 3 | 0
  Any Arthralgia, Across doses | 102
  Grade 3 Arthralgia, Across doses | 6
  Related Arthralgia, Across doses | 48
  Any Fatigue, Across doses | 165
  Grade 3 Fatigue, Across doses | 11
  Related Fatigue, Across doses | 72
  Any Fever, Across doses | 32
  Grade 3 Fever, Across doses | 1
  Related Fever, Across doses | 19
  Any Gastrointestinal, Across doses | 68
  Grade 3 Gastrointestinal, Across doses | 4
  Related Gastrointestinal, Across doses | 19
  Any Headache, Across doses | 127
  Grade 3 Headache, Across doses | 6
  Related Headache, Across doses | 47
  Any Myalgia, Across doses | 115
  Grade 3 Myalgia, Across doses | 7
  Related Myalgia, Across doses | 51
  Any Rash, Across doses | 17
  Grade 3 Rash, Across doses | 2
  Related Rash, Across doses | 8
  Any Urticaria, Across doses | 14
  Grade 3 Urticaria, Across doses | 1
  Related Urticaria, Across doses | 4

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3, Related and Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination. Grade 3 = event which prevented normal, everyday activities. Related = event assessed by the investigator as causally related to the study vaccination. Grade 3 and Related = grade 3 event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vacinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 596
Participants
  Any AE(s) | 20
  Grade 3 AE(s) | 3
  Related AE(s) | 2
  Grade 3 and Related AE(s) | 0

4. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade. Grade 3 SAE = SAE which prevented normal, everyday activities. Related SAE = SAE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 7)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 596
Participants
  Any SAE(s) | 4
  Grade 3 SAE(s) | 1
  Related SAE(s) | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: during the 30-day (Days 0-29) post-vaccination period; Serious adverse events: during the entire study period (from Day 0 up to Month 7).
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed. No related SAEs were reported and one (Uterine leiomyoma) was assessed as severe (Grade 3).
Arm/Group | Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/596
Serious Adverse Events (participants affected / at risk) | 4/596
Other Adverse Events (participants affected / at risk) | 443/596
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=596)
Bronchitis (Infections and infestations) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Mitral valve prolapse (Cardiac disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Typhoid fever (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=596)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 102 (149)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 168 (291)
Fatigue (General disorders) | 165 (258)
Gastrointestinal disorder (Gastrointestinal disorders) | 68 (93)
Headache (Nervous system disorders) | 127 (184)
Herpes zoster (Infections and infestations) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 115 (173)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 430 (922)
Polycystic ovaries (Reproductive system and breast disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 32 (42)
Rash (Skin and subcutaneous tissue disorders) | 17 (20)
Swelling (General disorders) | 119 (183)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7)
Urticaria (Skin and subcutaneous tissue disorders) | 14 (16)
Vaginitis bacterial (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.